CLINICAL TRIAL: NCT00445042
Title: A Phase II Study of Sorafenib in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Safety and Toxicity Study of Sorafenib in Patients With Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Bayer (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAC IRB#03-0194-05; Sorafenib-RCC-01
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: Metastatic Renal Cell Carcinoma; Metastatic RCC; Kidney Cancer; M3thodist
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Intrapatient dose escalation study of sorafenib
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — The initial dose of Sorafenib will be administered orally with a dose of 400 mg twice a day, daily. Intrapatient dose escalation will occur as defined in the protocol, providing no dose limiting toxicity (Grade 3 or 4) is observed.
  Other Names: Nexavar

SUMMARY:
The purpose of this study is to determine the safety and toxicity levels of Dose Escalated Sorafenib in the treatment of patients with renal cancer.

DETAILED DESCRIPTION:
Because tumors may have multiple mechanisms to induce angiogenesis, blockade with sorafenib may demonstrate efficacy. Doses of sorafenib (400 mg b.i.d.) as a single agent is with minimal toxicity, presents an opportunity to explore a more intensive drug administration. This study will allow individual patient titration (e,g,, intrapatient dose escalation) as per protocol.

This provides the basis for the dose escalation development of sorafenib. The study is designed to evaluate the ability for patients to dose escalate. Secondary endpoints include; response, time to progression, and overall survival in patients with MRCC. Tissue correlation to evaluate the impact of expression of receptor on clinical outcome will be retrospectively performed. Laboratory correlation of plasma VEGF levels will be correlated and evaluated to clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytological confirmed metastatic or unresectable clear cell renal cell carcinoma.
* No more than one prior systemic therapy. No prior vascular endothelial growth factor receptor agents.
* Patients with primary tumor in place are strongly encouraged to undergo nephrectomy prior to initiation of study agent.
* Prior palliative radiotherapy to metastatic lesion(s) is permitted.
* All major surgery of any type and/or radiotherapy must be completed at least 4 weeks prior to registration.
* Patients must have metastatic or unresectable disease.
* Paraffin RCC tissue blocks or unstained slides must be available.
* Karnofsky performance status > 70 % .
* Not pregnant
* Age > 18
* Must meet required initial laboratory values

Exclusion Criteria:

* No ongoing hemoptysis, or cerebrovascular accident within 12 months, or peripheral vascular disease with claudication on less than 1 block, or history of clinically significant bleeding.
* No deep vein thrombosis or pulmonary embolus within one year of study enrollment and no ongoing need for full-dose oral or parenteral anticoagulation. Low dose coumadin (1 mg) for maintenance of catheter patency or daily prophylactic aspirin is allowed.
* No evidence of current central nervous system (CNS) metastasis. All patients must undergo an MRI or CT scan of the brain (with contrast, if possible) within 42 days prior to registration. Any imaging abnormality indicative of CNS metastases will exclude the patient from the study.
* No significant cardiovascular disease defined as congestive heart failure (New York Heart Association Class II, II or IV) angina pectoris requiring nitrate therapy, or recent myocardial infarction (within the last 6 months).
* No patients with uncontrolled hypertension (defined as blood pressure of >160 mmHg systolic and/or > 90 mmHg diastolic on medication).
* Any ongoing requirement for systemic corticosteroid therapy is not permitted. Topical and/or inhaled steroids are allowed.
* No pre-existing thyroid abnormality whose thyroid function cannot be maintained in the normal range by medication are ineligible.
* No uncontrolled psychiatric disorder.
* Patients with delayed healing of wounds, ulcers and/or bone fractures are not eligible
* Patients with a 'currently active' second malignancy other than non-melanoma skin cancers are not eligible. Patients are not considered to have a 'currently active' malignancy if they have completed anti-cancer therapy and are considered by their physician to be a less than 30% risk of relapse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2005-11; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Tumor progression rate by RECIST criteria | restaging every 8 weeks

SECONDARY OUTCOMES:
Overall response rate | restaging every 8 weeks
Time to progression and overall survival | restaging every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — Baylor College of Medicine - Methodist Hospital
Locations (1):
- Methodist Hospital - Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No